CLINICAL TRIAL: NCT00005834
Title: A Phase III Trial of Dexamethasone, Cyclophosphamide, Etoposide, Cisplatin (DCEP) and G-CSF With or Without Thalidomide (NSC #66847) as Salvage Therapy for Patients With Refractory Multiple Myeloma
Brief Title: S9922 Combination Chemo Plus Filgrastim With or Without Thalidomide in Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S9922; S9922 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2000-06-02; First posted 2004-03-16 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cisplatin; Cyclophosphamide; Dexamethasone; Calcium Dobesilate; Etoposide; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chemo with thalidomide (Experimental): chemo with thalidomide
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: cyclophosphamide; Drug: dexamethasone; Drug: etoposide; Drug: thalidomide
- chemo without thalidomide (Active Comparator): chemo without thalidomide
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: cyclophosphamide; Drug: dexamethasone; Drug: etoposide

INTERVENTIONS:
Biological: filgrastim — Arms 1 and 2: 300 mcg (pts </= 60 kg) or 480 mcg (pts > 60 kg), SC beginning day 5
  Other Names: G-CSF
Drug: cisplatin — Arms 1 and 2: 15 mg/m2/d continuous IV days 1-4
  Other Names: platinol
Drug: cyclophosphamide — Arms 1 and 2: 400 mg/m2/d continuous IV days 1-4
  Other Names: cytoxan
Drug: dexamethasone — Arms 1 and 2: 40 mg/d PO days 1-4
  Other Names: decadron
Drug: etoposide — Arms 1 and 2: 40 mg/m2/d continuous IV days 1-4
  Other Names: VP-16
Drug: thalidomide — Arm 2: 800 mg/d (max dose) PO daily
  Other Names: thalomid
  Arms: chemo with thalidomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Thalidomide may stop the growth of tumor cells by stopping blood flow to the tumor. It is not yet known if combination chemotherapy is more effective with or without thalidomide for multiple myeloma.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without thalidomide in treating patients who have refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the overall and progression-free survival and remission rates in patients with refractory multiple myeloma treated with dexamethasone, cyclophosphamide, etoposide, cisplatin, and filgrastim (G-CSF) with or without thalidomide. II. Compare the qualitative and quantitative toxic effects of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior transplantation (yes vs no), prior treatment failure (resistant vs relapsing), prior treatment regimens (1-2 vs 3-4), and prior thalidomide (no vs some). Patients are randomized to one of two treatment arms. Arm I: Patients receive oral dexamethasone daily and cyclophosphamide, etoposide, and cisplatin (DCEP) IV continuously on days 1-4. Patients also receive filgrastim (G-CSF) subcutaneously daily beginning on day 5 and continuing until blood counts recover. Treatment continues every 3-4 weeks for 3 courses. Patients achieving stable disease or better proceed to maintenance chemotherapy with DCEP administered every 8 weeks for 3 additional courses. Arm II: Patients receive chemotherapy with DCEP as in arm I plus oral thalidomide daily. Thalidomide continues with maintenance chemotherapy and then continues after chemotherapy is completed until disease progression. Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 320 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage I, II, or III multiple myeloma with protein criteria present Quantifiable M-components of IgG, IgA, IgD, IgE AND/OR Urinary kappa or lambda light chain excretion No IgM peaks Quantifiable monoclonal proteins Received at least 1, but no more than 4 prior treatment regimens, including the following: Chemotherapy Bone marrow transplantation Biologic therapy Radiotherapy Interferon therapy or steroid pulsing given as maintenance therapy after transplantation or chemotherapy is not considered a separate treatment regimen Progressive disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 (3-4 allowed if due solely to bone pain) Life expectancy: At least 3 months Hematopoietic: Absolute granulocyte count at least 1,000/mm3 Platelet count at least 50,000/mm3 (at least 50% plasma cells in bone marrow) Hepatic: Bilirubin no greater than 2.5 times upper limit of normal (ULN) SGOT or SGPT no greater than 2.5 times ULN Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 60 mL/min Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use 2 methods of effective contraception for 4 weeks before, during, and for 4 weeks after study No other prior or concurrent malignancies within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or any other adequately treated stage I or II cancer in complete remission No grade 2 or greater preexisting peripheral neuropathy

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Prior thalidomide allowed if received less than 3 months of therapy Recovered from prior biologic therapy Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy and recovered No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics No concurrent hormonal therapy Radiotherapy: See Disease Characteristics At least 3 weeks since prior extensive or limited radiotherapy and recovered No concurrent radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2000-04; Primary Completion 2003-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
PFS | 18 months
  Length of time until progression - 25% increase from the baseline in myeloma protein production of other signs of disease progression such as hypercalcemia.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad A. Hussein, MD, Study Chair — The Cleveland Clinic
Locations (93):
- United States (93):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Hematology Oncology Associates, Atlantis, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington